CLINICAL TRIAL: NCT01867268
Title: Evaluating the Effect of Acetazolamide Administration and Prone Positioning Following Lumbosacral Spinal Surgery in Preventing Cerebro Spinal Fluid Leakage and Collection and Wound Dehiscence in Children.
Brief Title: Effect of Acetazolamide & Position in CSF Leakage and Collection and Wound Dehiscence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2137; 21843 (Other: Tehran University of Medical Sciences)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Fibrolipoma of Filum Terminale; Lipomyelomeningocele; Split Cord Malformation; Dermal Sinus; Tethered Cord Syndrome; Tumor
Keywords: Acetazolamide administration; prone positioning; Cerebrospinal fluid leakage; Cerebrospinal fluid collection; wound dehiscence
MeSH Terms: conditions — Lipomyelomeningocele; Neural Tube Defects; Spina Bifida Occulta; Neoplasms; Cerebrospinal Fluid Leak | interventions — Acetazolamide; Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acetazolamide (Experimental): administration of Acetazolamide for 10 days following the surgery
  Interventions: Drug: Acetazolamide
- Control (No Intervention): control group without any intervention
- Prone positioning (Experimental): Positioning the patient following surgery for 10 days
  Interventions: Other: prone positioning
- Acetazolamide and Prone positioning (Experimental): applying both Acetazolamide and prone positioning
  Interventions: Other: Acetazolamide+ prone positioning

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide administration for 10 days adjust dosage with weight of the patient
  Other Names: Diamox
  Arms: Acetazolamide
Other: prone positioning — prone positioning the patient for 10 days following the surgery
  Arms: Prone positioning
Other: Acetazolamide+ prone positioning — administration of acetazolamide and position the patient for 10 days following the surgery
  Arms: Acetazolamide and Prone positioning

SUMMARY:
* Purpose of study : to determine the preventive effect of acetazolamide administration, prone positioning, and the combination of both following the neurosurgical interventions in lumbosacral region for cerebrospinal fluid (CSF) leak, CSF collection and wound dehiscence.
* Sample size: 144
* intervention groups:

  * Group A: Acetazolamide administration for 10 days
  * Group B: prone positioning for 10 days
  * Group C: Acetazolamide administration and prone positioning for 10 days
  * Group D: no intervention
* Period of study: Autumn 2012 to the end of winter of 2015

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of Acetazolamide administration and prone positioning following lumbosacral spinal surgery in preventing cerebro-spinal fluid leakage and collection and wound dehissence in children admitted to Children Medical Center of Tehran since Autumn 2012 to the end of winter of 2015.The study is run under 4 categories of intervention:

* Group A: Acetazolamide administration for 10 days
* Group B: prone positioning for 10 days
* Group C: Acetazolamide administration and prone positioning for 10 days
* Group D: no intervention All patients are randomly assigned to these groups and when the patients faced with any of these complications, the protocol changes to Acetazolamide administration and prone positioning and the patient is considered as the failure of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Untethering surgery for primary tethered cord caused by thick filum
* Lipomyelomeningocele
* Split cord malformation management
* Untethering surgery in uncomplicated Dermal sinus
* Tumors needing intradural management in lumbosacral region
* Having any other disease with similar management technique

Exclusion Criteria:

* Infected dermoid tumors
* Intramedullary abscess
* Myelomeningocele surgery and related reoperation
* Meningocele
* Presence of hydrocephalus

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal fluid leakage | 1month
  leakage of CSF during 1 months following surgery
Cerebrospinal fluid collection | 1 month
  collection of the CSF beneath the skin during 1 month following the surgery
wound dehiscence | 1 month
  dehiscence of the surgical wound during the first month following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Farideh Nejat, MD, Study Director — Tehran University of Medical Sciences
Locations (1):
- Children'S Medical Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Chern JJ, Tubbs RS, Patel AJ, Gordon AS, Bandt SK, Smyth MD, Jea A, Oakes WJ. Preventing cerebrospinal fluid leak following transection of a tight filum terminale. J Neurosurg Pediatr. 2011 Jul;8(1):35-8. doi: 10.3171/2011.4.PEDS10502. PMID 21721886
- [Derived] Shahjouei S, Hanaei S, Habibi Z, Hoseini M, Ansari S, Nejat F. Randomized clinical trial of acetazolamide administration and/or prone positioning in mitigating wound complications following untethering surgeries. J Neurosurg Pediatr. 2016 Jun;17(6):659-66. doi: 10.3171/2015.8.PEDS15393. Epub 2016 Jan 29. PMID 26824595